CLINICAL TRIAL: NCT03557099
Title: A Multicentre, Open-label, Single-arm, Phase II Study to Evaluate the Safety and Efficacy of Hetrombopag Olamine in Patients With Severe Aplastic Anemia
Brief Title: A Study to Evaluate the Safety and Efficacy of Hetrombopag Olamine in Severe Aplastic Anemia （SAA） Patient
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-TPO-SAA-II
Record Dates: First submitted 2018-06-03; First posted 2018-06-14 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2020-04

CONDITIONS: Severe Aplastic Anemia
Keywords: SAA
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag Olamine (Experimental): Hetrombopag will be started at 7.5 mg/day and uptitrated according to the platelet count.
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — once daily

SUMMARY:
This is a Multicentre, Open-label, single-arm, Phase II Study to Evaluate the Safety and Efficacy of Hetrombopag Olamine in Patients With Severe Aplastic Anemia.

55 adult patients with SAA will be enrolled in the study. Treatment with Hetrombopag will be started at 7.5 mg/day and uptitrated according to the platelet count. The primary objective of the study is to assess the safety and efficacy of Hetrombopag in patients with SAA.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of refractory severe aplastic anemia, not meeting partial response criteria after at least one treatment course of immunosuppressive therapy, not suitable or unwilling to do hematopoietic stem cell transplantation.
2. Platelet count ≤ 30×109/L.
3. Signed informed consent.

Exclusion Criteria:

1. Bleeding and/or Infection not adequately responding to appropriate therapy.
2. Patients with a PNH clone size in neutrophils of ≥50%.
3. Treatment with immunosuppressive therapy within 6 months prior to study entry.
4. Any laboratory or clinical evidence for HIV infection. Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subjects screening.
5. ALT> 2.5 x upper limit of normal (ULN), AST> 2.5 x upper limit of normal (ULN) DBLI> 1.5 x upper limit of normal (ULN), Scr> upper limit of normal (ULN).
6. Subjects diagnosed with cirrhosis or portal hypertension.
7. Subjects diagnosed with tumor.
8. Patients with any prior history of congestive heart failure, arrhythmia, and peripheral arteriovenous thrombosis within 1 year. With a history of myocardial infarction or cerebral infarction within 3 months.
9. ECOG Performance Status of 3 or greater.
10. Female subjects who are nursing or pregnant within 6 months.
11. Subjects cannot take effective contraception.
12. Subjects have participated in other clinical trial within the 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects With Hematological Response | up to 18 weeks
  Hematological Response is defined by changes in the platelet count or platelet transfusion requirements, hemoglobin levels or number of red blood cell transfusions, neutrophil counts or G-CSF usage requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Peng G, He G, Chang H, Gao S, Liu X, Chen T, Li P, Han B, Miao M, Ge Z, Ge X, Li F, Li Y, Wang S, Wang Y, Shen Y, Zhang T, Zou J, Zhang F. A multicenter phase II study on the efficacy and safety of hetrombopag in patients with severe aplastic anemia refractory to immunosuppressive therapy. Ther Adv Hematol. 2022 Mar 30;13:20406207221085197. doi: 10.1177/20406207221085197. eCollection 2022. PMID 35371427